CLINICAL TRIAL: NCT00453856
Title: Efficacy of Sulfadoxine-Pyrimethamine in the Treatment of Symptomatic, Uncomplicated Plasmodium Falciparum Malaria Among 6-59 Month Old Children in Lambaréné
Brief Title: Efficacy of Sulfadoxine-Pyrimethamine for Treating Malaria in Gabonese Children
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated because of Early Treatment Failure in child.The justification for this decision are concerns about safety of children.
Sponsor: Albert Schweitzer Hospital, Netherlands (Unknown)
Collaborators: Albert Schweitzer Hospital (Other); Bill and Melinda Gates Foundation (Other)
Organization: Albert Schweitzer Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPTi-DRWG- SP Lambaréné
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2007-08-10 (Estimated); Status verified 2007-08

CONDITIONS: Malaria
Keywords: Malaria; Sulfadoxine; Pyrimethamine; Resistance; Gabon
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination

INTERVENTIONS:
Drug: Sulfadoxine Pyrimethamine

SUMMARY:
IPTi, a strategy whereby infants are provided treatment doses of antimalarials at routine vaccination visits, has been shown to significantly reduce malaria and anemia in two studies in Tanzania. However the results obtained in Gabon are not similar. Many factors are likely to influence the efficacy or effectiveness IPTi. It is reasonable to assume that the efficacy of IPTi will be influenced markedly by the sensitivity of Plasmodium falciparum to the antimalarial drug (Sulfadoxine-Pyrimethamine) used for IPTi.

In order to interpret the results of individual IPTi trials conducted by the IPTi Consortium, and to provide information for policy makers regarding the predicted efficacy of IPTi, it is essential to obtain information on antimalarial drug sensitivity of Sulfadoxine-Pyrimethamine now that the IPTi trial has been conducted. The simplest and most universally accepted measure of testing for antimalarial drug efficacy is the "in vivo efficacy study," which follows a standardized World Health Organization protocol.

A second reason for evaluating drug resistance as an adjunct to the IPTi trials is to determine if the intervention increases the carriage and/or spread of drug resistant P. falciparum parasites.

Thirdly the overall effect at the community level of selection of resistant genotypes in IPTi-recipients is unclear.

DETAILED DESCRIPTION:
Administration of standard single oral dose of sulfadoxine-pyrimethamine to children aged 6-59 month old children in Lambaréné at enrolment, if eligible according to the approved protocol.

139 subjects will be enrolled and treated with Sulfadoxine-Pyrimethamine for uncomplicated malaria. Thereafter each subject will be followed according to the approved protocol

The proportion of subjects with Adequate Clinical and Parasitological response (ACPR) by day 28, Early Treatment Failure (ETF), Late Clinical Failure (LCF) and Late Parasitological Failure (LPF)will be evaluated.

secondly the frequency of molecular markers for Sulfadoxine-Pyrimethamine drug resistance will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients
* Aged 6 to 59 months
* Body weight between 7.5 to 30 kg
* uncomplicated falciparum malaria with parasitaemia between 1,000/µL and 200,000/µL
* Ability to tolerate oral therapy
* Informed consent, oral agreement of the child if appropriate

Exclusion Criteria:

* Still in IPTi trial and/or still in any other intervention trial
* Known G6PD-deficiency
* Presence of severe malnutrition
* Inability to drink or breastfeed
* Recent history of convulsions, lethargy or unconsciousness;
* Signs of severe and complicated
* Mixed/mono infection that includes a non-P. falciparum species.
* Hb < 7g/dl
* Inability to attend stipulated follow-up visits.
* History of hypersensitivity reactions to the drug being evaluated

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 139 (Estimated)
Dates: Start 2007-03

PRIMARY OUTCOMES:
Measure the clinical and parasitological efficacy of SP among patients aged between 6-59 months suffering from uncomplicated P falciparum malaria,

SECONDARY OUTCOMES:
Determine the frequency of molecular markers for drug resistance

CONTACTS AND LOCATIONS:
Overall Officials: Martin P Grobusch, MD, Study Director — Medical Research Unit, Albert Schweitzer Hospital Lambaréné; Saadou Issifou, MD MSc, Principal Investigator — Albert Schweitzer Hospital
Locations (1):
- Medical Research Unit of the Albert Schweitzer Hospital, Lambaréné, Moyen-Ogooué Province, Gabon

REFERENCES:
- [Derived] Mombo-Ngoma G, Oyakhirome S, Ord R, Gabor JJ, Greutelaers KC, Profanter K, Greutelaers B, Kurth F, Lell B, Kun JF, Issifou S, Roper C, Kremsner PG, Grobusch MP. High prevalence of dhfr triple mutant and correlation with high rates of sulphadoxine-pyrimethamine treatment failures in vivo in Gabonese children. Malar J. 2011 May 14;10:123. doi: 10.1186/1475-2875-10-123. PMID 21569596
- See also: (Homepage of the Medical Research Unit, Lambaréné) — http://www.lambarene.org